CLINICAL TRIAL: NCT01351818
Title: The Fayds Project: Adipocyte Function and Somtropin Deficiency
Brief Title: Adipocyte Function and Somtropin Deficiency
Acronym: FAYDS
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring SAU (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Other Study IDs: FER-SOM-2004-01
Record Dates: First submitted 2011-05-02; First posted 2011-05-11 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Growth hormone: Patients with a condition
  Interventions: Drug: Growth Hormone

INTERVENTIONS:
Drug: Growth Hormone

SUMMARY:
To assess the influence of exogenous GH (growth hormone) administration on adipocyte endocrine function (leptin, adiponectin, and resistin) and on ghrelin secretion in children with delayed growth due to GH deficiency.

Study hypothesis: hormones produced by the adipocyte (leptin, adiponectin, and resistin) and ghrelin may exert a certain control on production of GH and IGF-I, and GH may in turn have a regulatory effect on such hormones.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes aged from 5 to 12 years, Tanner stage 1, with no signs of imminent pubertal development. Amenable to treatment with recombinant somatropin in the approved indication of low growth due to GH deficiency
* Selection of recombinant somatropin by the physician in the treatment authorization request, and subsequent approval of such treatment by the relevant growth hormone committee
* Body Mass Index (BMI) within ±1 SD

Exclusion Criteria:

* Children with any of the reported contraindications for treatment with recombinant somatropin, existence of active neoplasms, progression or recurrence of intracranial lesion, etc. will not be studied
* Diabetes mellitus
* Intestinal inflammatory disease
* Celiac disease
* Uncontrolled hyperthyroidism
* AIDS
* Other diseases causing chronic malabsorption, hypercatabolism or malnutrition conditions
* Chronic liver disease
* Eating disorders: anorexia, bulimia, etc
* Long-term treatment with anti-obesity drugs or drugs causing malabsorption

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with GH deficiency
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2005-05; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the potential influence of exogenous GH administration on adipocyte endocrine function (leptin, adiponectin, and resistin) and on ghrelin secretion | 1 year

SECONDARY OUTCOMES:
Height assessment (using Harpenden stadiometer) | 1 year
Weight assessment | 1 year
BMI assessment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (12):
- Spain (12):
  - Investigational site, Badajoz, Badajoz
  - Investigational site, Don Benito, Badajoz
  - Investigational site, Cáceres, Cáceres
  - Investigational site, Cadiz, Cádiz
  - Investigational site, Córdoba, Córdoba
  - Investigational site, Granada, Granada
  - Investigational site, Huelva, Huelva
  - Investigational site, Jaén, Jaen
  - Investigational site, Murcia, Murcia
  - Investigational site, Málaga, Málaga
  - Investigational site, Seville, Sevilla
  - Investigational site, Santa Cruz de Tenerife, Tenerife